CLINICAL TRIAL: NCT01724385
Title: Intravitreal Bevacizumab for Proliferative Diabetic Retinopathy With New Dense Vitreous Hemorrhage After Full Panretinal Photocoagulation
Brief Title: Intravitreal Bevacizumab for Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Yosanan Yospaiboon, Professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I55116
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Vitreous Hemorrhage; Proliferative Diabetic Retinopathy
Keywords: bevacizumab,; proliferative diabetic retinopathy,; vitreous hemorrhage,
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intravitreal bevacizumab injection (Experimental): intravitreal injection of bevacizumab 1.25 mg
  Interventions: Drug: intravitreal injection of bevacizumab

INTERVENTIONS:
Drug: intravitreal injection of bevacizumab — intravitreal injection of bevacizumab
  Other Names: Avastin

SUMMARY:
To evaluate the efficacy of intravitreal bevacizumab injections for treatment of proliferative diabetic retinopathy (PDR) with new dense vitreous hemorrhage (VH) after previous full panretinal photocoagulation (PRP).

DETAILED DESCRIPTION:
The investigators will carry out a prospective study in patients with PDR and prior complete laser treatment who presented with new dense VH. All eyes will be treated with intravitreal injection of bevacizumab (1.25 mg). Complete ophthalmic examination and/or ocular ultrasonography will be performed at baseline and 1, 6, 12 weeks and 6, 9, 12 months after first injection. Re-injection will be done in non-clearing and recurrent VH.

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetes mellitus
* proliferative diabetic retinopathy
* prior complete panretinal photocoagulation
* presented with new dense vitreous hemorrhage

Exclusion Criteria:

* one-eyed patient
* previous intraocular surgery
* severe lens opacity precluding fundus examination
* advance glaucoma
* history of thromboembolic events such as myocardial infarction and cerebrovascular accident
* uncontrolled systemic hypertension, systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg
* known coagulation abnormalities or current use of anticoagulant medications other than aspirin
* known allergies to any relevant drugs in this study
* evidence of external ocular infection such as conjunctivitis and significant blepharitis.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The percentage of eyes that vitreous hemorrhage has been completely resolved | 12 months
  The patients with PDR and prior complete laser treatment who presented with new dense VH. All eyes were treated with intravitreal bevacizumab injection. Complete ophthalmic examination and/or ocular ultrasonography were performed at baseline and 1, 6, 12 weeks and 6, 9, 12 months after first injection.

SECONDARY OUTCOMES:
The change in best corrected visual acuity (BCVA) from baseline | 12 months
  The best corrected visual acuity (BCVA) was performed at baseline and 1, 6, 12 weeks and 6, 9, 12 months after first injection.

OTHER OUTCOMES:
Numbers of injection | 12 months
  Numbers of intravitreous bevacizumab injection in a 12-month period

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Sinawat, M.D., Principal Investigator — Department of Ophthalmology, Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand